CLINICAL TRIAL: NCT01412567
Title: Comparison of Recombinant Hepatitis B Vaccine Plus Hepatitis B Immune Globulin (HBIG) Versus Vaccine Plus Placebo for Prophylaxis of Hepatitis B Infection in Newborns of Hepatitis B Surface Antigen (HBsAg) Positive Mothers
Brief Title: Vaccine+HBIG Versus Vaccine+Placebo for Newborns of HBsAg+ Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Collaborators: Indian Council of Medical Research (Other Government); Lady Hardinge Medical College (Other Government)
Responsible Party: Prof Shiv Kumar Sarin, G B Pant Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: LHMC-1
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; HBsAg; Antenatal; Pregnancy; Vertical transmission; Placenta; HBV DNA
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccine+HBIG (Active Comparator)
  Interventions: Drug: Vaccine+HBIG
- Vaccine+Placebo (Placebo Comparator)
  Interventions: Drug: Vaccine+Placebo

INTERVENTIONS:
Drug: Vaccine+HBIG — Recombinant hepatitis B vaccine at birth, 6 weeks, 10 weeks, and 14 weeks in the dose of 10 mcg (0.5 mL), by intramuscular injection in the anterolateral thigh; PLUS HBIG in the dose of 0.5 mL intramuscularly immediately after birth
  Arms: Vaccine+HBIG
Drug: Vaccine+Placebo — Recombinant hepatitis B vaccine at birth, 6 weeks, 10 weeks, and 14 weeks in the dose of 10 mcg (0.5 mL), by intramuscular injection in the anterolateral thigh; PLUS placebo intramuscularly immediately after birth
  Arms: Vaccine+Placebo

SUMMARY:
Prevention of perinatal transmission is essential to decrease the global burden of chronic HBV. Recombinant HBV vaccine and hepatitis B immunoglobulin (HBIG) given after delivery to the newborns of HBsAg positive mothers is the standard of care for prevention of HBV in babies. Some studies have however, shown that vaccine alone may be equally effective. Hence, immunoprophylaxis with hepatitis B vaccine with or without HBIG is effective in prevention of transmission of overt HBV infection to the babies. The primary outcome measure of most of the trials on immunoprophylaxis was the occurrence of hepatitis B, defined as a blood specimen positive for hepatitis B surface antigen (HBsAg). However, whether this immunoprophylaxis also prevents HBsAg negative HBV infection (occult HBV infection) in babies is not known. In the present study the investigators evaluated the efficacy of the two regimens; vaccination alone and compared it with vaccination plus HBIG administration at birth in preventing transmission of both overt and occult HBV infection to the newborn babies.

ELIGIBILITY:
Inclusion Criteria:

* Newborn babies of mothers who were found to be HBsAg positive

Exclusion Criteria:

* Babies of mothers who had any symptoms of liver disease during the pregnancy such as jaundice, pruritus, ascites, or gastrointestinal bleed;
* Babies of mothers taking anti-viral treatment during pregnancy;
* Babies of mother with pregnancy related complications; and
* Babies of mothers who refused to participate in the study.

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 259 (Actual)
Dates: Start 2005-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
remaining free of any HBV infection (either overt or occult) plus development of adequate immune response to vaccine at 18 weeks of age | 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Pande C, Sarin SK, Patra S, Kumar A, Mishra S, Srivastava S, Bhutia K, Gupta E, Mukhopadhyay CK, Dutta AK, Trivedi SS. Hepatitis B vaccination with or without hepatitis B immunoglobulin at birth to babies born of HBsAg-positive mothers prevents overt HBV transmission but may not prevent occult HBV infection in babies: a randomized controlled trial. J Viral Hepat. 2013 Nov;20(11):801-10. doi: 10.1111/jvh.12102. Epub 2013 Apr 23. PMID 24168259